CLINICAL TRIAL: NCT06050031
Title: Level of DNA-fragmentation Before and After Antioxidant-based Therapies in Male Infertility: An Observational Study on Factors Influencing the Treatment Effects
Brief Title: Level of DNA-fragmentation Before and After Antioxidant-based Therapies in Male Infertility
Status: Not yet recruiting | Type: Observational
Sponsor: Janna Pape (Other)
Responsible Party: Sponsor-Investigator, Janna Pape, Principal Investigator, Dr. med. Janna Pape, Universitätsklinik fur Frauenheilkunde, Inselspital Bern
Organization: Universitätsklinik fur Frauenheilkunde, Inselspital Bern (Other)
Other Study IDs: 2023-00611
Record Dates: First submitted 2023-09-11; First posted 2023-09-22 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Infertility, Male
Keywords: antioxidant; DNA-fragmentation; Oxidation-reduction potential; Lifestyle
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: Intake of antioxidant supplement — All participants will supplent oral antioxidants (individual or combined which can be obtained without prescription, and which are not regulated as a pharmaceutical drug) over three months.

SUMMARY:
The investigators will investigate the effect of antioxidants and lifestyle factors on the level of oxidative stress. As oxidative stress cannot be directly measured, it will be approximated by the DNA fragmentation index (DFI) which reflects the level of DNA damage in sperm caused by oxidative stress.

DETAILED DESCRIPTION:
This is a one-site prospective exploratory study at the University Clinic for Gynaecological Endocrinology and Reproductive Medicine in Bern. On total 78 men with male infertility will be recruited.

The primary objective of the study is to assess the effectiveness of 3 months of antioxidant-based therapy on changing patients' DFI level.

The objective of the study is to assess the effect of 3 months of antioxidant-based therapy on the level of DFI. We are primarily interested in testing whether the treatment effectiveness (i.e. the change in DFI level) depends on the initial level (i.e. before treatment) and treatment adherence.

The data will be collected by the physicians and added to the REDcap study registry. Access to the total data set is only permitted for the principal investigator.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate
* Written consent
* Men with infertility problems who want to start an infertility treatment with their partner

Exclusion Criteria:

* No measurement of DNA fragmentation possible
* Intake of prescribed medications
* Exposure to toxins
* Chronic diseases

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — No, it is based on the biological gender.
Study Population: Male patients with infertility
Sampling Method: Non-Probability Sample
Enrollment: 78 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
DFI | At baseline and after three months of antioxidant-treatment
  DNA-fragmentation measured by sperm-chromatin-structure-assay (SCSA)

SECONDARY OUTCOMES:
Sperm concentration | At baseline and after three months of antioxidant-treatment
  Sperm concentration [10^6/mL]
Sperm motility | At baseline and after three months of antioxidant-treatment
  Total sperm progressive motility [%] Oxidation-reduction potential [mV/10-6 sperm/mL]
Oxidation-reduction potential in ejaculate | At baseline and after three months of antioxidant-treatment
  Oxidation-reduction potential [mV/10-6 sperm/mL]
Alcohol consumption | At baseline and during the three months of antioxidant-treatment
  Alcohol consumption [unit per week]
BMI | At baseline and after the three months of antioxidant-treatment
  BMI [kg/m2]
Smoking | At baseline and during the three months of antioxidant-treatment
  Cigarette consumption [number of cigarettes per week]
Treatment adherence | During three months of antioxidants
  Averaged missing capsules per week (100%, 75%, 50%, 25%) during treatment
Implantation rate | 10-12 days after timed intercourse, insemination or embryo transfer in the first treatment cycle after the antioxidant treatment
  Endocrine pregnancy by measuring hCG in blood sample on day 10-12 after timed intercourse, insemination or embryo transfer
Clinical pregnancy rate | 5 weeks after timed intercourse, insemination or embryo transfer in the first treatment cycle after the antioxidant treatment
  Clinical pregnancy confirmed by ultrasound, 5 weeks after timed intercourse, insemination or embryo transfer
Live birth rate | 9 months after timed intercourse, insemination or embryo transfer in the first treatment cycle after the antioxidant treatment
  Birth of a living baby nine months after timed intercourse, insemination or embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Michael von Wolff, Prof, Study Chair — Universitätsklinik fur Frauenheilkunde, Inselspital Bern

IPD SHARING:
Plan to Share IPD: No